CLINICAL TRIAL: NCT00837850
Title: A Randomised Prospective Trial of SmartSet HV and Palacos R Bone Cements in Primary Total Hip Arthroplasty. A Radiostereometric Analysis of the Charnley Femoral Component.
Brief Title: SmartSet HV and Palacos R RSA Bone Cements in Primary Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 094-02
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Arthritis
Keywords: total hip arthroplasty; Charnley stem; RSA; non-inflammatory arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Device: Bone cement 1
- 2 (Active Comparator)
  Interventions: Device: Bone cement 2

INTERVENTIONS:
Device: Bone cement 1 — Bone cement SmartSet® HV
  Other Names: SmartSet HV
  Arms: 1
Device: Bone cement 2 — Bone cement Palacos R
  Other Names: Palacos R
  Arms: 2

SUMMARY:
A randomised radiostereometric study comparing SmartSet HV and Palacos R acrylic bone cements.

DETAILED DESCRIPTION:
The fixation of components in total hip arthroplasty has a significant effect on the long-term survival of the prostheses. Bone cement in total joint replacement acts as an anchoring medium for the prosthesis and provides a barrier to the ingress of wear debris into bone surfaces. However, there are significant differences in cement behaviour among differing types of cement. A clinical study based on the Norwegian Arthroplasty Register demonstrated that there is an increased rate of revision due to aseptic loosening of femoral components implanted with low-viscosity cement compared with that of high-viscosity.

Studies have shown that high early migration for certain designs of femoral prosthesis can be a predictor for clinical loosening. RSA is a technique enabling calculation of the three-dimensional translational and rotational movements of the implant relative to the bone, and therefore provides an ideal technique to detect early micromotion of implants.

ELIGIBILITY:
Inclusion Criteria:

* patients in need for total hip arthroplasty

Exclusion Criteria:

* patients with an existing condition such as malignancy, pregnancy, severe osteoporosis and disabling musculoskeletal problems (other than in the hips),
* patients on corticosteroid treatment,
* patients who had already participated in a clinical study with an investigational product in the last 6 months.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2002-10; Primary Completion 2003-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Distal migration of the charnley femoral stem | 2010

SECONDARY OUTCOMES:
Rotational movements of the charnley femoral stem | 2010

CONTACTS AND LOCATIONS:
Overall Officials: Otto S. Husby, PhD, Principal Investigator — St.Olavs hospital HF

REFERENCES:
- [Result] Husby OS, Haugan K, Benum P, Foss OA. A prospective randomised radiostereometric analysis trial of SmartSet HV and Palacos R bone cements in primary total hip arthroplasty. J Orthop Traumatol. 2010 Mar;11(1):29-35. doi: 10.1007/s10195-010-0087-x. Epub 2010 Mar 3. PMID 20198403